CLINICAL TRIAL: NCT04945707
Title: A Double-blind,Randomized, Placebo-controlled Study to Assess Exercise Tolerance After Iron Repletion With Ferric Derisomaltose (Monoferric®) IV Compared to Placebo in Heart Failure With Preserved Ejection Fraction and With Iron Deficiency.
Brief Title: Impact of Intravenous Iron Repletion On Mechanisms of Exercise InTolerance in HFpEF (IRONMET-HFpEF)
Acronym: IRONMETHFpEF
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pharmacosmos A/S (Industry); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Gregory D. Lewis, M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P001501; R01HL151841 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-30 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Iron-deficiency; Heart Failure With Preserved Ejection Fraction
Keywords: Heart Failure with Preserved Ejection Fraction; Iron Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferric derisomaltose; Saline Solution

STUDY DESIGN:
Intervention Model Description: This is a double-blind, prospective, randomized, placebo-controlled study to assess exercise tolerance after iron repletion with a single dose of ferric derisomaltose (Monoferric®) IV compared to placebo in heart failure with preserved ejection fraction and with iron deficiency. Randomization will be stratified by sex and will be performed in permutated blocks of 4 to assure balanced group sizes
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded staff (clinical research nurse and unblinded investigator) prepare and administer study drug to subject and document and follow safety events. The subject is blinded. A tented covering will allow adequate viewing of the IV site, but outside of the view of the subject. All blinded staff will not be present during study drug infusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): Ferric derisomaltose (Monoferric®) 1000 mg X 1 (for subject <50 kg, 20 mg/kg X1)
  Interventions: Drug: Ferric Derisomaltose 1000 Mg in 100 mL INTRAVENOUS SOLUTION [Monoferric]
- Arm 2 (Placebo Comparator): Normal Saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric Derisomaltose 1000 Mg in 100 mL INTRAVENOUS SOLUTION [Monoferric] — Ferric derisomaltose (Monoferric) 1000 mg X1 (for subject <50 kg, 20 mg/kg
  Other Names: Monoferric
  Arms: Arm 1
Drug: Placebo — Normal saline
  Other Names: Normal Saline
  Arms: Arm 2

SUMMARY:
The primary objective of this study is to determine if the correction of functional iron deficiency by administering a single dose of intravenous iron (ferric derimaltose or Monoferric®) in participants with heart failure with preserved ejection fraction (HFpEF) will improve exercise capacity as measured by the change in peak oxygen uptake (peak VO2) from baseline to 12 weeks.

DETAILED DESCRIPTION:
A double-blind, prospective, randomized, placebo-controlled study to assess change in exercise capacity after iron repletion with a single dose of ferric derisomaltose (Monoferric®) IV compared to placebo in heart failure with preserved ejection fraction and with functional iron deficiency.

Sixty-six HFpEF participants who have functional iron deficiency will be recruited from the Cardiopulmonary Exercise Testing (CPET) Laboratory and will have a recent or scheduled clinical care CPET with exercise hemodynamic assessment. These measurements will serve as baseline measures. After undergoing other baseline measurements such as echocardiogram, actigraphy, research biomarkers, and the Kansas City Cardiomyopathy Questionnaire (KCCQ) participants will be randomized (2:1) to either a single dose of ferric derisomaltose (Monoferric®)1000 mg/100 ml (n=44) or placebo (n=22).

Given that the iron drug formulation is of brown color and the placebo is clear, unblinded staff members will be assigned to order, pick up and administer drug to the subject. The subject is blinded; therefore, the drug will be infused using a tented covering over the arm in which the IV has been placed. The tented covering will allow adequate viewing of the IV site, but outside of the view of the subject. All blinded staff will not be present during study drug infusion. Prior to infusion the subject will undergo vital signs; blood pressure, heart rate, and temperature. A peripheral intravenous catheter will be placed followed by an infusion of Monoferric 1000 mg (for subjects less than 50 kg, 20 mg/kg) as per current FDA-approved dosing or placebo over 20 minutes. Vital signs will be performed immediately after dosing and after 30 minutes. Subjects will remain in the clinic for observation for 30 minutes following infusion.

Randomization will be stratified by sex and will be performed in permutated blocks of 4 to assure balanced group sizes. In order to allocate without bias, and in a manner blinded to both participants and investigators, we will use random number generation at the time of randomization.

Participants will return for a CPET, echocardiogram, actigraphy, KCCQ, ECG, complete metabolic panel, and blood draw for research biomarkers, cardiovascular exam, and assessment of adverse experiences. A subset of subjects (n=33) will undergo a CPET with exercise hemodynamic assessment. The remaining subjects will undergo an noninvasive CPET (N=33)

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age) able to provide informed consent.
2. Stable heart failure (NYHA II-IV) for at least 4 weeks
3. Heart Failure with Preserved left ventricular ejection fraction.(Left ventricular ejection fraction ≥ 50 % obtained within 6 months of informed consent.
4. NT-proBNP ≥ 125 pg/mL without ongoing atrial fibrillation/flutter. If ongoing atrial fibrillation/flutter at the time of sample collection, NT-proBNP must be ≥ 250 pg/mL OR patients must have a history of pulmonary capillary wedge pressure ≥ 15 mm Hg during rest or the slope of pulmonary capillary wedge pressure to cardiac output (PCWP/CO) ≥ 2.0 mmHg/L/min during upright exercise (Eisman et al., Circ Heart Fail. 2018 May;11(5):e004750.).OR subjects must have a heart failure hospitalization within the last 12 months prior to screening OR Chronic diastolic dysfunction on echocardiography as evidenced by: Left Atrial Enlargement (LAE): LA diameter ≥ 3.8cm in women, ≥ 4.0 cm in men or LA length ≥ 5.0 cm or LA area ≥ 20 cm2 OR LA volume ≥ 55mL or LA volume index ≥ 29ml/m2 or Left Ventricular Hypertrophy (LVH): septal thickness or posterior wall thickness ≥ 1.1 cm OR For patients in sinus rhythm: E/e' ratio ≥15 at septal annulus, or E/e' ratio ³13 at lateral annulus, or average E/e' ratio ³14. For patients in atrial fibrillation: E/e' ≥ 11 at the septal annulus.
5. Hemoglobin >9.0 g/dL AND <15.0 g/dL .
6. Serum ferritin <100 ng/mL OR 100 to 300 ng/mL with TSAT <20%, but NOT ferritin < 15 ng/mL.
7. Demonstrate diminished exercise capacity: ≤ 75 % predicted peak VO2 as determined by a Cardiopulmonary Exercise Test (CPET) at the time of screening
8. Perform a maximal effort CPET by achieving a Respiratory Exchange Ratio (RER) of ≥ 1.05

Exclusion Criteria:

1. Current or planned intravenous iron supplementation. Iron-containing multivitamins (<30 mgs /day) are permitted.
2. Known hypersensitivity reaction to any component of ferric derisomaltose (Monofer®)
3. History of acquired iron overload (e.g. hemochromatosis), or the recent receipt (within 3 months) of erythropoietin stimulating agent, IV iron therapy, or blood transfusion.
4. Documented active gastrointestinal bleeding
5. Anemia with known cause other than iron deficiency or chronic disease
6. Acute myocardial infarction, acute coronary syndrome, transient ischemic attack, or stroke within 3 months of enrollment.

7 Presence of any condition that precludes exercise testing such as:

a. Claudication that limits exertion b. Uncontrolled bradyarrhythmia or tachyarrhythmia (according to Investigator judgment, pacemaker treatment is allowed as long as the same pacing mode/activity can be used at baseline and follow-up CPET) c. Clinically significant musculoskeletal disease or orthopedic conditions that limit the ability to perform the CPET (e.g., arthritis or injury in the foot, leg, knee or hip) d. Severe obesity (BMI > 50.0 kg/m2) e. Any other non-heart failure condition that, in the opinion of the Investigator, that is the primary limitation to exercise. 8. Severe renal dysfunction (eGFR< 20 ml/min/1.73m2) 9. Severe liver disease (ALT or AST > 3x upper limit of normal, alkaline phosphatase or bilirubin >2x upper limit of normal) 10. Active malignancy other than non-melanoma skin cancers 11. Female participant of child-bearing potential who is pregnant, lactating, or not willing to use adequate contraceptive precautions during the study and for up to 5 days after the last scheduled dose of study medication.

12. Planned surgical procedure during the trial period 13. Inability to return for follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-11-26 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The change in peak oxygen uptake (peak VO2) from baseline to week 12 in HFpEF subjects with functional iron deficiency following a single dose of ferric derisomaltose or placebo. | 12 weeks
  Peak VO2 measured by a maximal effort Cardiopulmonary Exercise Test (CPET)

SECONDARY OUTCOMES:
Change in resting pulmonary capillary wedge pressure (PCWP) | Baseline to week 12
  Measured by right heart catheterization with CPET
Change in resting pulmonary artery pressure (PAP) | Baseline to week 12
  Measured by right heart catheterization with CPET
Change in exercise pulmonary capillary wedge pressure/ cardiac output slope (PCWP/CO slope) | Baseline to week 12
  Measured by right heart catheterization with CPET
Change in exercise pulmonary arterial pressure/ cardiac output slope (PAP/CO slope) | Baseline to week 12
  Measured by right heart catheterization with CPET
Change in exercise peripheral oxygen extraction C(a-v)O2 | Baseline to week 12
  Measured by right heart catheterization with CPET
Change in resting and exercise pulmonary vascular resistance (PVR) | Baseline to week 12
  Measured by right heart catheterization with CPET
Change in hepcidin | Baseline and week 12
  Measured in blood samples
Change in transferrin saturation to hepcidin ratio | Baseline and week 12
  Measured in blood samples
Change in hemojuvelin | Baseline and week 12
  Measured in blood samples
Change in soluble transferrin receptor level | Baseline and week 12
  Measured in blood samples
Change in NTpBNP | Baseline and week 12
  Measured in blood samples
Change in C-reactive Protein | Baseline and week 12
  Measured in blood samples
Change in physical activity level as measured by accelerometer motion-sensing data collection | Baseline to week 12
  Measured by Actigraphy
Change in Quality of Life | Baseline to week 12
  Measured by Kansas City Cardiomyopathy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Greg Lewis, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lewis GD, Malhotra R, Hernandez AF, McNulty SE, Smith A, Felker GM, Tang WHW, LaRue SJ, Redfield MM, Semigran MJ, Givertz MM, Van Buren P, Whellan D, Anstrom KJ, Shah MR, Desvigne-Nickens P, Butler J, Braunwald E; NHLBI Heart Failure Clinical Research Network. Effect of Oral Iron Repletion on Exercise Capacity in Patients With Heart Failure With Reduced Ejection Fraction and Iron Deficiency: The IRONOUT HF Randomized Clinical Trial. JAMA. 2017 May 16;317(19):1958-1966. doi: 10.1001/jama.2017.5427. PMID 28510680
- [Background] Houstis NE, Eisman AS, Pappagianopoulos PP, Wooster L, Bailey CS, Wagner PD, Lewis GD. Exercise Intolerance in Heart Failure With Preserved Ejection Fraction: Diagnosing and Ranking Its Causes Using Personalized O2 Pathway Analysis. Circulation. 2018 Jan 9;137(2):148-161. doi: 10.1161/CIRCULATIONAHA.117.029058. Epub 2017 Oct 9. PMID 28993402